CLINICAL TRIAL: NCT06604078
Title: Elucidating the Impact of Social Wellness and Artificial Intelligence on the Psychological Consequences of Breast Cancer Imaging
Brief Title: Breast Cancer AI Imaging Study
Status: Completed | Type: Observational
Sponsor: University of Central Florida (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00005494
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer; Breast Cancer Screening
Keywords: Breast Cancer; Artifical Inteligence; AI
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study aims to develop a social health platform called MammoChat (https://MammoChat.com) that allows patients to share their real-world patient data to a trusted network for development of clinical intelligence to improve patient outcomes. Therefore:

1. The investigator will establish a Discourse social network where patients can anonymously and securely share their breast imaging and interact with other patients.
2. The investigator will use standardized questionnaires to understand the impact of use of the social network on outcomes related to breast cancer screening such as anxiety.
3. The investigator will assemble a crowdsourced, de-identified radiographic repository for training, testing, and validating AI models aimed at earlier and more accurate disease detection for breast cancer.

DETAILED DESCRIPTION:
With over 40,000,000 mammograms run annually in the US, there are psychological consequences of breast cancer imaging that are well documented among patients such as stress and anxiety from largely false positive or indeterminant readings by radiologists.

This UCF MammoChat platform is one of the first projects that engages patients to donate their breast cancer imaging in an effort to reduce the psychological consequences of breast cancer imaging using social networks and artificial intelligence.

This repository will be supported and maintained by the University of Central Florida College of Medicine (UCF COM) Clinical and Aerospace Research team. These clinical research coordinators will operate the repository, including administering patients, imaging sites and transfers through an administrative panel.

ELIGIBILITY:
Inclusion Criteria:

* Adults, ages 18 and older
* Had a radiographic breast cancer imaging test, either for screening or diagnosis of breast cancer, with either positive or negative results performed in a US institution.
* Have an email account with access to a reliable internet connection or smartphone

Exclusion Criteria:

* Minors , ages under 18
* Prisoners. Given the repository design, prisoners are unlikely to participate and provide a consent
* Adults who are unable to provide consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be enrolled online from across the US.
  Potential participants will not be screened for eligibility. In the informed consent process, participants will self-disclose if they have done breast cancer imaging at a US institution.
  Pregnant women may choose to participate in the repository.
Sampling Method: Non-Probability Sample
Enrollment: 199 (Actual)
Dates: Start 2024-09-05 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
AI Model Development | 25 years
  Train, test and validate AI models with de-identified radiographic images collected from participants.
Psychological Impact of Breast Cancer Screening | 25 years
  Assess user anxiety using the standardized COS-BC (Consequences of Screening in Breast Cancer) questionnaire.
Social Discourse for Patients on Wellness Network | 25 years
  Assess patient participation on Discourse social network using standardized user metrics such as activity logs, images posted, other interactions, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Dexter Hadley, M.D., PhD, M.S.E, Principal Investigator — University of Central Florida
Locations (1):
- University of Central Florida, Orlando, Florida, United States